CLINICAL TRIAL: NCT00638664
Title: Optimized MRI Evaluation of Maximal Temporal and Spatial Measurability of the Cardiac Chambers and Thoracic Great Vessels. A Comparison of MR Acquisition Pulse Sequences.
Brief Title: Evaluation of the MRI in Measuring the Cardiac Chambers and Thoracic Great Vessels
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, David Feiglin, Chairman of Radiology Department, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 3149
Record Dates: First submitted 2008-02-01; First posted 2008-03-19 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Chambers
Keywords: conventional pulse sequences for MR; cardiac chambers and walls; cardio-thoracic vasculature; the great vessels; coronary vasculature; cardiac; great vessels

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We are seeking volunteers to participate in a research study to determine the optimal imaging parameters for visualization of the heart and its great vessels so that errors in computer data analysis is minimized and clinical accuracy is maximized.

Participation in this study will involve having an MRI of the heart. This study will allow us to determine the ability to measure the volumes of your heart chambers in both the left and right side of your heart without using any aggressive (invasive) technique or the use of ionizing radiation (x-rays or gamma rays). The study will also allow us to measure changes in the cardiac chamber volumes during the cardiac cycle and determine whether this can be done rapidly and accurately. The study will also allow us to determine whether this technique can be used for routine clinical use.

DETAILED DESCRIPTION:
The ability to obtain accurate cyclical functional information of the cardiac chambers plays a continuing important clinical diagnostic role in the evaluation and monitoring of patients with a wide range of cardiac pathologies, including those embarking on or continuing cardiotoxic chemotherapeutic regimes, as well as patients with lung disease.

The current imaging modalities used for non-invasive imaging of the heart include echocardiography and radionuclide ventriculography. Echocardiographic evaluation of cardiac function is primarily limited to the left ventricle and functional measurements are based on volumetric estimates in turn based usually on geometric assumptions. That is, the volume calculation is based on a limited number of non orthogonal linear measurements assuming a regular (non complex) chamber morphology. This study technique provides no biologic hazard to the patient.

Radionuclide ventriculography does allow for 3D cardiac data acquisition and theoretical evaluation of biventricular function. However, the technique does not provide the same degree of spatial resolution that echocardiography can provide. Radionuclide ventriculography is a commonly accepted diagnostic procedure but does involve use of ionizing radiation.

Magnetic Resonance imaging techniques (of the heart) allows relatively high resolution cross sectional imaging. For example a 512X512 matrix over a 40cm field of view provides in plane resolution better that 1mm. No assumptions are made in regard chamber cross sectional area and hence volume morphology. The slice thickness is determined in advance and may be in the range of 1-10mm. MR data ca be acquired sequentially throughout the cardiac cycle and thus provide a time varying 3D map of the cardiac chambers and related structures during the cardiac cycle.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* Able to understand and sign consent without surrogate signature
* Subject weight is within the 300lb limit of the MR scanning table
* Subject's bodily habitus allows the subject to fit within the MR bore
* Subject being able to lie quiescent for a period of up to 60 minutes in a supine position
* Subject would be able to hold breath at times for periods of 15-30 seconds

Exclusion Criteria:

* Subjects with pacemakers, TENS units, metallic prostheses, metal foreign bodies such as bullets, shrapnel, metallic slivers, shavings or foreign bodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology Clinic Center Watch Website
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 1995-05 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Feiglin, MD, Principal Investigator — SUNY Upstate MU
Locations (1):
- University Radiology Associates, Syracuse, New York, United States